CLINICAL TRIAL: NCT01187680
Title: Polyethylene Glycol Adhesion Barrier Reduces Adhesions After Gynecologic Laparoscopy; a Prospective Randomized Controlled Pilot Study
Brief Title: Efficacy of Sprayable PEG Barrier in Gynecologic Laparoscopy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Financial and organisational reasons
Sponsor: Radboud University Medical Center (Other)
Collaborators: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: E. Bakkum, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RU-RTB-0002
Record Dates: First submitted 2010-07-19; First posted 2010-08-24 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-08

CONDITIONS: Postoperative Adhesion; Peritoneal Adhesion, Nos
Keywords: Tissue adhesions; Laparoscopy
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spraygel (Experimental)
  Interventions: Device: Spraygel
- Control (Active Comparator)
  Interventions: Device: Control

INTERVENTIONS:
Device: Spraygel
  Arms: Spraygel
Device: Control — Good surgical technique, no adhesion barrier
  Arms: Control

SUMMARY:
The purpose of the study is to investigate whether sprayable PEG barrier is effective in reducing adhesions in laparoscopic gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Undergoing gynecologic laparoscopy

Exclusion Criteria:

* Suspected malignancy
* Incomplete adhesiolysis during initial laparoscopy
* Pregnancy
* Lactating
* Stage IV endometriosis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2002-10; Primary Completion 2004-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
successful adhesion prevention
  Adhesion prevention was defined as successful if no de novo fromed adhesion were found at second look laparoscopy.

SECONDARY OUTCOMES:
LABS adhesion score
Adhesion sites
  Reduction in the number of sites covered with adhesions

CONTACTS AND LOCATIONS:
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands